CLINICAL TRIAL: NCT06029283
Title: Effect on Oral-cardio Health From Dietary Nitrate Loaded Functional Gum
Brief Title: Dietary Nitrate Functional Gum Effect on Gingivitis and Heart Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Harlan Shiau, Clinical associate professor / program director, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HP-00106795
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Gingivitis; Cardiovascular Diseases; Gingival Diseases; Gingival Bleeding; Periodontal Diseases
Keywords: gingivitis; dietary nitrate; periodontal disease
MeSH Terms: conditions — Gingivitis; Cardiovascular Diseases; Gingival Diseases; Gingival Hemorrhage; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo arm of non-dietary nitrate gum (Placebo Comparator): Placebo gum with no dietary nitrate
  Interventions: Other: Placebo chewing gum
- Test arm of dietary nitrate containing gum (Experimental): Functional gum with dietary nitrate
  Interventions: Dietary Supplement: dietary nitrate

INTERVENTIONS:
Dietary Supplement: dietary nitrate — dietary nitrate in a chewing gum delivery vehicle
  Arms: Test arm of dietary nitrate containing gum
Other: Placebo chewing gum — placebo chewing gum
  Arms: Placebo arm of non-dietary nitrate gum

SUMMARY:
The purpose of this research is to determine the effects of a chewing gum containing dietary nitrate to gingival and heart health. Dietary nitrates are commonly found in leafy vegetables and beets. The information learned from the study may help further understand the interconnection of oral health and heart health. The study is looking for individuals who present with mild to moderate gum irritation or bleeding.

In the study participants will be randomized into either a group that will use a chewing gum containing dietary nitrate, or use a placebo chewing gum during a three-week period.

Participants in the study will have a simple gingival exam, x-rays if needed, and small samples of saliva and blood collected. All participants will also undergo a routine tooth cleaning. Participants will be asked to breathe in a tube to sample the levels of nitric oxide. Finally, participants will have their heart health measured with a device that is like a blood pressure cuff.

DETAILED DESCRIPTION:
The purpose of the project is to characterize, in subjects with gingival inflammation, the effect of a prebiotic dietary nitrate formulated chewing gum on the oral microbiome. In order to assess this, gingival health and parameters related to vascular health are observed:

The study is testing the hypothesize that short term use of functional gum will have improved inflammatory measures of the gingiva and beneficial cardiovascular impact. The study hopes to discover if any observed changes to oral and cardiovascular measures may be associated to changes to oral microbiome composition.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with mild to moderate gingivitis, defined with a MGI score of at least 2.0
* Subjects must have a minimum of 20 natural teeth
* Subjects must be able to chew gum

Exclusion Criteria:

* Significant alveolar bone loss (>3.0 mm CEJ to bone)
* Requirement for antibiotic pre-medication prior to dental procedures
* Systemic antibiotic use in past 14 days to current.
* Use of anti-inflammatory (NSAIDs) or in past 14 days
* Use of anticoagulant therapy or in past 14 days.
* Current smokers
* Pregnancy
* Use of any oral rinses such as, but not limited to chlorhexidine, essential oils, cetylpyridinium chloride during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Gingival inflammation | 0 and 21 days
  Gingival index or similar data collected.
Microbiome profile | 0 and 21 days
  salivary sample collected
Blood vessel elasticity | 0 and 21 days
  CV profiler device used
nitric oxide | 0 and 21 days
  Breathalyzer type test

CONTACTS AND LOCATIONS:
Overall Officials: Harlan Shiau, Principal Investigator — Clinical Assoc. Prof.
Locations (1):
- University of Maryland School of Dentistry, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No